CLINICAL TRIAL: NCT05869786
Title: Investigation of the Effect of Virtual Reality-Mediated Rehabilitation on Upper Extremity Functions in Ischemic Stroke Patients
Brief Title: The Effect of Virtual Reality-Mediated Rehabilitation in Ischemic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ahmet Kivanc Menekseoglu, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023.04.43
Record Dates: First submitted 2023-04-18; First posted 2023-05-22 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hemiplegia
MeSH Terms: conditions — Hemiplegia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This prospective, randomized and controlled study will be conducted with patients diagnosed with stroke. Among the patients who are admitted to outpatient or inpatient rehabilitation program in SBU Kanuni Sultan Süleyman PTR clinic, 30 patients diagnosed with stroke who meet the inclusion criteria will be included in the study. Patients diagnosed with stroke will be randomized into two groups using a computer program (Virtual reality group, control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Virtual Reality Group (Experimental): Participants in both groups will receive a conventional rehabilitation program. Participants in the virtual reality group will receive virtual reality-mediated upper extremity rehabilitation for 3 weeks, 5 sessions per week, each session lasting 30 minutes (450 minutes in total). In the virtual reality intervention, participants will be asked to control the games with hand, wrist and forearm movements in front of a computer screen in front of the SensoRehab® sensor that can detect hand movements through gloves. 3 different games will be intervened for 10 minutes each, totaling 30 minutes per day.
  Interventions: Device: Virtual Reality Mediated Upper Extremity Rehabilitation (SensoRehab®); Other: conventional rehabilitation program
- Control Group (Active Comparator): Participants in the control group will be instructed in hand, finger, wrist and forearm therapeutic exercises by a physiotherapist. Participants in both groups will receive a conventional rehabilitation program.
  Interventions: Other: conventional rehabilitation program; Behavioral: Exercise

INTERVENTIONS:
Device: Virtual Reality Mediated Upper Extremity Rehabilitation (SensoRehab®) — In the virtual reality intervention, participants will be asked to control the games with hand, wrist and forearm movements in front of a computer screen in front of the SensoRehab® sensor that can detect hand movements through gloves.
  Arms: Virtual Reality Group
Other: conventional rehabilitation program — conventional rehabilitation program
Behavioral: Exercise — Participants in the control group will be instructed in hand, finger, wrist and forearm therapeutic exercises by a physiotherapist.
  Arms: Control Group

SUMMARY:
The aim of the study was to investigate the effectiveness of virtual reality-mediated upper extremity rehabilitation added to the conventional rehabilitation program on upper extremity, quality of life, range of motion and spasticity in patients with stroke.

DETAILED DESCRIPTION:
This prospective, randomized and controlled study will be conducted with patients diagnosed with stroke. Among the patients who are admitted to outpatient or inpatient rehabilitation program in SBU Kanuni Sultan Süleyman PMR clinic, 30 patients diagnosed with stroke who meet the inclusion criteria will be included in the study. Patients diagnosed with stroke will be randomized into two groups using a computer program (Virtual reality group, control group). Participants in both groups will receive a conventional rehabilitation program. Participants in the virtual reality group will receive virtual reality-mediated upper extremity rehabilitation for 3 weeks, 5 sessions per week, each session lasting 30 minutes (total 450 minutes). In the virtual reality intervention, participants will be asked to control the games with hand, wrist and forearm movements in front of a computer screen in front of the SensoRehab® sensor that can detect hand movements through gloves. 3 different games will be intervened for 10 minutes each, totaling 30 minutes per day.

Participants in the control group will be instructed in hand, finger, wrist and forearm therapeutic exercises by a physiotherapist.

After the intervention, patients will be evaluated in terms of upper extremity functions, quality of life, range of motion and spasticity.

All evaluations will be repeated before, after and 3 months after the intervention. Routine 3-month PMR outpatient clinic control is recommended for patients with stroke. Therefore, no additional hospital visit is requested from the patients due to the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age,
* History of Ischemic Stroke
* Accept to participate in the study,

Exclusion Criteria:

* Presence of known central nervous system or peripheral nervous system disease other than stroke, presence of progressive neurologic deficit,
* Uncontrolled hypertension, diabetes, cardiovascular disease etc.
* Cognitive impairment causing difficulty in executing simple commands
* Epilepsy
* Botulinum toxin application to the upper extremity in the last 6 months
* Change in the medical treatment used for spasticity in the last 6 months
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer upper extremity scale | Change from Baseline Fugl-Meyer upper extremity scale at 3rd Month After Intervention
  This scale is a stroke-specific, performance-based scale and each parameter is scored as 0; unsuccessful, 1; partially successful and 2; completely successful performance. This scale consists of five sections: motor function, balance, sensation, range of motion and pain. The motor function assessment section is scored as 100 points (66 upper extremities and 34 lower extremities), sensation (light touch and position sense) 24 points, balance (6 sitting and 8 standing) 14 points, range of motion 44 points and joint pain 44 points.

SECONDARY OUTCOMES:
Functional Independence Measure | Change from Baseline Functional Independence Measure at 3rd Month After Intervention
  Participants' functional status will be assessed by Functional Independence Measure. In this scale, the functional status of patients is evaluated with 18 questions under 6 sub-headings, each question is scored between 1-7. Higher scores indicate better functional status.
Handgrip Strength | Change from Baseline Handgrip Strength at 3rd Month After Intervention
  The handgrip strength of the participants will be evaluated with a dynamometer.
Modified Ashworth Scale | Change from Baseline Modified Ashworth Scale at 3rd Month After Intervention
  Upper extremity muscle spasticity of the participants will be evaluated with the modified Ashworth Scale. According to this scale, spasticity is evaluated between 0-4. Higher points mean more spasticity.
Stroke Impact Scale | Change from Baseline Stroke Impact Scale. at 3rd Month After Intervention
  The quality of life of the participants will be evaluated with the Stroke Impact Scale.It consists of 8 subsections and 59 questions. Each question is scored by rating the difficulty experienced in the last week on a 5-point scale. The score for each section ranges from 0-100. Higher scores are associated with better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: AHmet Kivanc Menekseoglu, MD, Principal Investigator — Kanuni Sultan Suleyman Research and Training Hospital
Locations (1):
- Ahmet Kıvanç Menekşeoğlu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No